CLINICAL TRIAL: NCT03260166
Title: An Open-label Study for Assessing the Efficacy and Safety of Nicotinamide Treatment for Lupus-associated Skin Lesions in Patients With Cutaneous Lupus Erythematosus or Systemic Lupus Erythematosus
Brief Title: Nicotinamide Treatment for Lupus-associated Skin Lesions in Lupus Erythematosus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Hunan Provincial Natural Science Foundation of China (Unknown); National Key Clinical Specialty Construction Project of China (Unknown)
Responsible Party: Principal Investigator, Qianjin Lu, MD, PhD, Professor and Director, Dept. of Dermatology, The Second Xiangya Hospital of Central South University, Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFK201707
Record Dates: First submitted 2017-08-10; First posted 2017-08-24 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Cutaneous Lupus Erythematosus; Systemic Lupus Erythematosus Rash
Keywords: nicotinamide; lupus-associated skin lesion; lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous | interventions — Niacinamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- nicotinamide (Experimental): Patients will receive 10 nicotinamide tablets orally twice daily (nicotinamide 500 mg, p.o., Bid) for a period of 3 months. Each tablet contains 50 mg of nicotinamide.
  Interventions: Drug: nicotinamide

INTERVENTIONS:
Drug: nicotinamide — Drug: nicotinamide; Pharmaceutical form: tablet; Route of administration: oral
  Other Names: Niacinamide

SUMMARY:
This clinical study will test the efficacy and safety of nicotinamide for lupus-associated skin lesions refractory to the treatment of hydroxychloroquine plus low-dose corticosteroids in patients with cutaneous lupus erythematosus (CLE) or systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
Backgrounds: Lupus erythematosus (LE) is an autoimmune disease affecting various organs. Lupus-associated skin lesions are the dominant clinical manifestations of cutaneous lupus erythematosus (CLE) and also occur in 70%~80% of patients with systemic lupus erythematosus (SLE), and usually involve the sunlight-exposure sites such as the face, neck and hands, which affects the personal appearance dramatically and causes substantial psychological impact to the patients.

While antimalarials such as hydroxychloroquine (HCQ) have been widely used as a first-line treatment for lupus-associated skin lesions, 30% of patients with lupus do not respond to this medication. Other available therapies such as corticosteroids and thalidomide can also be applied, however, their toxic side effects limit the clinical use. Recent studies by the investigators have shown that nicotinamide, a water-soluble vitamin whose side effects are considered as minimal, can protect MRL/lpr mice (a lupus-like mouse model) from skin lesions and autoantibody production. Thus it is hypothesized that nicotinamide treatment could be a novel therapy for lupus-associated skin lesions in patients with LE.

Design of Study: This is a single center, uncontrolled, open-label study to assess the efficacy and safety of nicotinamide for lupus-associated skin lesions refractory to the treatment of HCQ plus low-dose corticosteroids in patients with CLE or SLE.

Methods: For CLE or SLE patients with lupus-associated skin lesions scoring >=4 on the Revised Cutaneous Lupus Erythematosus Disease Area and Severity Index (RCLASI) that have been refractory to the treatment of HCQ plus low-dose corticosteroids (<=0.5 mg/kg/d) during the past two months, oral nicotinamide (500 mg twice daily) will be given consecutively for 3 months while the current regimen including HCQ and corticosteroids be maintained without change. The end points include clinical response and immunological changes, as well as safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 18 years and 65 years.
2. Patients clinically and histopathologically diagnosed as cutaneous lupus erythematosus (CLE) that have not respond to treatment with hydroxychloroquine (200-400 mg/day) plus corticosteroids at a dosage less than the equivalent of 0.5mg/kg/day of prednisone for the preceding two months or a longer period.
3. Patients diagnosed as SLE (meeting the 1997 American College of Rheumatology criteria for SLE) that present with lupus-associated skin lesions that have not respond to treatment with hydroxychloroquine (200-400 mg/day) plus corticosteroids at a dosage less than the equivalent of 0.5mg/kg/day of prednisone for the preceding two months or a longer period.
4. Revised Cutaneous Lupus Erythematosus Disease Area and Severity Index (RCLASI) ≥4; for patients with SLE, Safety of Estrogens in Lupus Erythematosus National Assessment version of the systemic lupus erythematosus disease activity index (SELENA-SLEDAI) is within the range between 0 and 9.
5. Written informed consent form.

Exclusion Criteria:

1. Severe comorbidities including heart failure (≥grade III NYHA), respiratory failure, renal insufficiency (creatinine clearance ≤30 ml/min), hepatic insuf¬ficiency (alanine aminotransferase or aspartate aminotransferase ≥2 times of the upper limit of the normal range), or active severe neuropsychiatric manifestations of SLE.
2. Acute severe infection such as sepsis and cellulitis, or a history of infection of hepatitis B or C virus, Mycobacterium tuberculosis, or human immunodeficiency virus (HIV).
3. A history of treatment with nicotinamide, niacin, or multi-vitamins in the recent month.
4. A history of treatment with rituximab or other biologics; or a history of treatment with high-dose corticosteroids (≥1.5 mg/kg/d), immunosuppressants, tripterygium glycosides, or intravenous immunoglobin G (IVIG) in the preceding three months.
5. Patients not suitable for using nicotinamide due to comorbidities including pruritic skin diseases such as atopic dermatitis and urticaria, vertigo, dizziness, headache, hyperglycemia, and hyperuricemia; patients not suitable for using hydroxychloroquine due to conditions including retinopathy or hypersensitivity to hydroxychloroquine.
6. Patients with drug abuse, alcohol abuse, or mental disorders that are unable to cooperate or adhere to treatment.
7. Pregnancy or lac¬tation in females.
8. Participants in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
A change in Revised Cutaneous Lupus Erythematosus Disease Area and Severity Index (RCLASI) activity score | from baseline (at visit 0) to 3 months treatment (at visit 3)
  The higher the RCLASI score, the worse of the lupus-associated skin lesion is.

SECONDARY OUTCOMES:
A change in RCLASI activity score | from baseline (at visit 0) to 1, 2, 4, and 6 months treatment (at visit 1, 2, 4, and 5), respectively
  The higher the RCLASI score, the worse of the lupus-associated skin lesion is.
Response Rate and Remarkable Response Rate at 1, 2, 3, 4, and 6 months, respectively | 1 month, 2 months, 3 months, 4 months, and 6 months
  Response is defined as a ≥ 4-point reduction or a ≥20% reduction in RCALSI activity score. Remarkable Response is defined as a ≥50% reduction in RCALSI activity score.
Number of Relapses | 4 months, 6 months
  Relapse means that if the patient's RCLASI activity score has a ≥ 4-point reduction or a ≥20% reduction than at baseline during the 3-month treatment, and then the RCLASI activity score increase to be no lower than at baseline after stopping using nicotinamide in the following 3 months.
A change in Dermatology Life Quality Index (DLQI) score | from baseline (at visit 0) to 1 month, 2 months, 3 months, 4 months, and 6 months (at visit 1, 2, 3, 4, and 5), respectively
  DLQI reflect the quality of life related to skin manifestations.
A change in Physician's Global Assessment (PGA) score | from baseline (at visit 0) to 1 month, 2 months, 3 months, 4 months, and 6 months (at visit 1, 2, 3, 4, and 5), respectively
A change in the percentage of different T helper cell (Th) subsets among CD4+ T lymphocytes | from baseline (at visit 0) to 1 month, 2 months, 3 months, 4 months, and 6 months (at visit 1, 2, 3, 4, and 5), respectively
  At each time point, the percentage of Th1, Th2, Th17, regulatory T cell (Treg), and follicular helper T cell (Tfh) subsets among CD4+ T lymphocytes in peripheral venous blood of the patient will be measured by flow cytometry. 5 ml of peripheral venous blood will be collected from the patient at each time point, of which 4.5 ml will be used in this flow cytometry assay.
A change in the serum level of cytokines interferon (IFN)γ, interleukin (IL)-4, IL-17A, transforming growth factor (TGF)-β, IL-10, IL-21, and IL-6 | from baseline (at visit 0) to 1 month, 2 months, 3 months, 4 months, and 6 months (at visit 1, 2, 3, 4, and 5), respectively
  At each time point, the serum level of cytokines IFNγ, IL-4, IL-17A, TGF-β, IL-10, IL-21, and IL-6 in the patient's venous blood will be measured using enzyme linked immunosorbent assay (ELISA) or Bio-Plex methods. 5 ml of peripheral venous blood will be collected from the patient at each time point, of which 0.5 ml will be used in this ELISA or Bio-Plex assay.
A change in serum levels of complement 3 (C3), C4, and C1q | from baseline (at visit 0) to 1 month, 2 months, 3 months, 4 months, and 6 months (at visit 1, 2, 3, 4, and 5), respectively
  This is for evaluation of the potential effects of nicotinamide on serum levels of complements that are associated with lupus activity
A change in the results of urine sediment test | 1 month, 2 months, 3 months, 4 months, and 6 months
  This is for evaluation of the potential effects of nicotinamide on renal damage.
Dose reduction of concomitant corticosteroids | from baseline (at visit 0) to 3 months, 4 months, and 6 months (at visit 3, 4, and 5), respectively
A change in SELENA-SLEDAI (Safety of Estrogens in Lupus Erythematosus National Assessment version of the systemic lupus erythematosus disease activity index) | from baseline (at visit 0) to 1 month, 2 months, 3 months, 4 months, and 6 months (at visit 1, 2, 3, 4, and 5), respectively
  This outcome is only evaluated for patients with SLE.
A change in British Isles Lupus Assessment Group 2004 Index (BILAG-2004) | from baseline (at visit 0) to 1 month, 2 months, 3 months, 4 months, and 6 months (at visit 1, 2, 3, 4, and 5), respectively
  This outcome is only evaluated for patients with SLE.
Incidence of side effects | 3 months
  Possible side effects of nicotinamide include flushing and itching of the skin, cardiac arrhythmia, dizziness, nausea, epigastric discomfort, loss of appetite, elevated blood glucose, and elevated blood uric acid. The major side effects of HCQ that need to be monitored include retina toxicity.
Incidence of side effects | 6 months
  Possible side effects of nicotinamide include flushing and itching of the skin, cardiac arrhythmia, dizziness, nausea, epigastric discomfort, loss of appetite, elevated blood glucose, and elevated blood uric acid. The major side effects of HCQ that need to be monitored include retina toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Qianjin Lu, MD, PhD, Principal Investigator — Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No